CLINICAL TRIAL: NCT03033199
Title: A Multi-center Randomized Clinical Trial of Regulating Gut Microbiota by Probiotic Agents in Management of Immune Thrombocytopenia
Brief Title: Clinical Trial of Gut Microbiota in the Management of Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Jinan Central Hospital (Other); The Second Hospital of Shandong University (Other); Qianfoshan Hospital (Other); Qingdao University (Other); Yantai Yuhuangding Hospital (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITP-Microbiota
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Immune Thrombocytopenia
Keywords: Gut microbiota; Immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic Agent Combining HD-DXM (Active Comparator): probiotic capsules containing three viable and freezedried strains-Lactobacillus acidophilus,Lactobacillus casei, and Bifidobacterium bifidum：2 capsules, bid x 4 weeks for one cycle. It will be given for one or two cycles.
  Dexamethasone 40mg per day, 4 consecutive day
  Interventions: Drug: Probiotic Agent; Drug: Dexamethasone
- HD-DXM (Active Comparator): Dexamethasone 40 mg per day, 4 consecutive days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Probiotic Agent — probiotic capsules containing three viable and freezedried strains-Lactobacillus acidophilus,Lactobacillus casei, and Bifidobacterium bifidum：2 capsules, bid x 4 weeks for one cycle. It will be given for one or two cycles.
  Arms: Probiotic Agent Combining HD-DXM
Drug: Dexamethasone — Dexamethasone 40 mg per day, 4 consecutive days

SUMMARY:
Primary immune thrombocytopenia (ITP) is an acquired autoimmune bleeding disorder, accounting for about 1/3 of clinical hemorrhagic diseases. Loss of immune tolerance leading to increased platelet destruction and decreased platelet production is the main pathogenesis of ITP. Dysbiosis of the gut microbiota was found in many autoimmune diseases like rheumatic arthritis(RA),inflammatory bowel disease(IBD),multiple sclerosis and probiotic treatment or fecal microbiota transplantation(FMT) which can regulate the gut microbiota has good clinical efficacy in those disorders. One ITP patient with ulcerative colitis(UC) was treated with FMT and got progressive but significant increase in platelet level and lasted for several years.

DETAILED DESCRIPTION:
The investigators are undertaking a multicenter, single-arm study of 60 primary ITP adult patients from 5 medical centers in China. All the participants are randomly divided into two groups to orally intake either probiotic supplements (n = 30) or placebo (n = 30) for 4 weeks in addition with high dose dexamethasone(40 mg/d for 4 days). Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* need of treatment(s) (including, but not limited to, low dose of corticosteroids) to minimize the risk of clinically significant bleeding. Need of on-demand or adjunctive therapy alone does not qualify the patient as refractory
* primary ITP confirmed by excluding other supervened causes of thrombocytopenia

Exclusion Criteria:

* pregnancy
* hypertension
* cardiovascular disease
* diabetes
* liver and kidney function impairment
* HCV, HIV, HBsAg seropositive status
* patients with systemic lupus erythematosus and/or antiphospholipid syndrome
* patients with known gastro-intestinal bleeding.
* use of antibiotics, prebiotics or probiotics in the past 4 weeks;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Platelet count | From date of randomization until the date of first documented progression,up to 12 months
  R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Shandong University Qilu hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang Y, Cai Y, Zhang X, Kong X, Su J. Altered gut microbiota in RA: implications for treatment. Z Rheumatol. 2017 Jun;76(5):451-457. doi: 10.1007/s00393-016-0237-5. PMID 27909795
- [Background] Vaghef-Mehrabany E, Alipour B, Homayouni-Rad A, Sharif SK, Asghari-Jafarabadi M, Zavvari S. Probiotic supplementation improves inflammatory status in patients with rheumatoid arthritis. Nutrition. 2014 Apr;30(4):430-5. doi: 10.1016/j.nut.2013.09.007. Epub 2013 Dec 17. PMID 24355439
- [Background] Smits LP, Bouter KE, de Vos WM, Borody TJ, Nieuwdorp M. Therapeutic potential of fecal microbiota transplantation. Gastroenterology. 2013 Nov;145(5):946-53. doi: 10.1053/j.gastro.2013.08.058. Epub 2013 Sep 7. PMID 24018052
- [Background] Zamani B, Golkar HR, Farshbaf S, Emadi-Baygi M, Tajabadi-Ebrahimi M, Jafari P, Akhavan R, Taghizadeh M, Memarzadeh MR, Asemi Z. Clinical and metabolic response to probiotic supplementation in patients with rheumatoid arthritis: a randomized, double-blind, placebo-controlled trial. Int J Rheum Dis. 2016 Sep;19(9):869-79. doi: 10.1111/1756-185X.12888. Epub 2016 May 2. PMID 27135916